CLINICAL TRIAL: NCT02888600
Title: Stress Management Training for Healthy Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Collaborators: University of Pittsburgh (Other); Virginia Commonwealth University (Other)
Responsible Party: Principal Investigator, David Creswell, Professor, Carnegie Mellon University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1R01AT008685-01 (NIH)
Record Dates: First submitted 2016-08-15; First posted 2016-09-05 (Estimated); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Psychological Stress; Loneliness
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness Training (Active Comparator): The Mindfulness Meditation Program consists of eight weekly 2- 2.5 hour group sessions, a day-long retreat in the sixth week, and daily mindfulness meditation homework.
  Interventions: Behavioral: Mindfulness Training
- Health Education (Active Comparator): The Health Education Program also consists of eight weekly 2- 2.5 hour group sessions, a day-long retreat in the sixth week, and daily health practice homework
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Mindfulness Training — Guided mindfulness meditation and stress management training
  Arms: Mindfulness Training
Behavioral: Health Education — Guided health education and stress management training
  Arms: Health Education

SUMMARY:
This study is a two-arm randomized controlled trial comparing two 8-week stress management programs for reducing inflammation and improving well-being among older adults.

DETAILED DESCRIPTION:
A growing body of literature has demonstrated how stress can affect social relationships, health, and well-being during the aging process. Here, the investigators will test how two different programs can be used to facilitate healthy aging by helping individuals manage stress. One program will teach participants mindfulness meditation techniques while the other will educate participants about how to manage their health.

N=188 older adults will visit the study's central laboratory for a baseline visit and complete several days of daily experience sampling before being randomized into one of the two 8-week stress management programs. Participants will complete several days of daily experience sampling at the midpoint and conclusion of the intervention before returning to a study site to complete a follow-up assessment at both 1-week and 3-months after the end of the program.

This project will provide important information about how each training program can be used to promote well-being, health, and better social functioning in older adults. This work will ultimately inform the design of more efficacious and efficient stress-management interventions to facilitate healthy aging.

ELIGIBILITY:
Inclusion Criteria:

* English speaking

Exclusion Criteria:

* [Exclusion criteria are masked from public viewing until data collection is complete. Please contact project managers.]

Ages: 65 Years to 93 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 190 (Actual)
Dates: Start 2016-06-28 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-11-29 (Actual)

PRIMARY OUTCOMES:
Circulating markers of inflammation, Interleukin-6 and C Reactive Protein | Change from baseline to 1-week post-intervention and 3-month follow-up
  Measured via blood samples

SECONDARY OUTCOMES:
Pro-inflammatory gene expression | Change from baseline to 1-week post-intervention
Self-reported relational distress | Change from Baseline to Intervention Weeks 4 and 8
  Evaluated using ecological momentary assessment
Self-reported loneliness | Change from baseline to 1-week post-intervention and 3-month follow-up
  Evaluated using UCLA loneliness scale and ecological momentary assessment
Self-reported awareness of experiences and reactivity to experience during resting state | 1-week post-intervention and 3-month follow-up
  Questionnaire assessing the frequency in which participants notice a variety of positive, neutral, and negative experiences and their reactivity to those experiences during a 5-minute resting state period
Working memory in daily living | Change from baseline to intervention weeks 4 and 8
  Assessed via a dot memory ambulatory smartphone-based task administered at six timepoints per day, for three days in a row, at baseline and at Intervention weeks 4 and 8
Implicit acceptance of self | 1-week post-intervention and 3-month follow-up
  Assessed via an Implicit Association Test (IAT) behaviorally quantifying the association between self and acceptance/judgment

OTHER OUTCOMES:
Health practices | Change from baseline to 1-week post-intervention and 3-month follow-up
  Evaluated by questionnaires asking about diet, caffeine consumption, alcohol use, stress reduction, exercise, recreational drug use, cold or flu, flu shots
Mental health | Change from baseline to 1-week post-intervention and 3-month follow-up
  Evaluated using Beck Depression Inventory
Self-reported stress | Change from baseline to 1-week post-intervention and 3-month follow-up
Mindfulness | Change from baseline to 1-week post-intervention and 3-month follow-up
  Evaluated using Mindful Attention Awareness Scale
Connectedness to nature | Change from baseline to 1-week post-intervention and 3-month follow-up
  Evaluated using Nature Connection Scale
Personality | Change from baseline to 1-week post-intervention and 3-month follow-up
  Evaluated using NEO Personality Inventory
Social network and social support | Change from baseline to 1-week post-intervention and 3-month follow-up
  Evaluated using Social Network Index and Interpersonal Support Evaluation List
Self-reported psychological distress | Change from baseline to 1-week post-intervention and 3-month follow-up
Trait affect | Change from baseline to 1-week post-intervention and 3-month follow-up
  Evaluated using Stanford Measure of Actual, Ideal, and Avoided Affect
Trait hostility | Change from baseline to 1-week post-intervention and 3-month follow-up
  Evaluated using Cook-Medley Hostility Scale
Attachment style | Change from baseline to 1-week post-intervention and 3-month follow-up
  Evaluated using Adult Attachment Scale
Attitudes towards aging | Change from baseline to 1-week post-intervention and 3-month follow-up
  Evaluated using Attitudes to Aging Questionnaire
Immune functioning | Change from baseline to 1-week post-intervention and 3-month follow-up
  Assessed via stimulated IL-6 production and glucocorticoid resistance
Cellular aging | Change from baseline to 1-week post-intervention and 3-month follow-up
  Assessed via telomeres and telomerase
Markers of inflammation | Assessed at 3-month follow-up only
  Assessed via hair sample
Social interaction quality and quantity | Change from Baseline to Intervention Weeks 4 and 8
  Assessed via ecological momentary assessment
Self-reported psychological distress | Change from Baseline to Intervention Weeks 4 and 8
  Assessed via ecological momentary assessment
Home practice quality and quantity | Assessed daily throughout the eight-week intervention period
  Assessed by self-reported practice length, enjoyment of practice, usefulness of practice, trouble concentrating, mental fatigue, stress, and irritation during practice.
Treatment expectations | Assessed prior to beginning of intervention, during Intervention Weeks 4 and 8
  Assessed by optimism about treatment and expectations for treatment outcome,
Instructor and class ratings | Assessed prior to beginning of intervention, during Intervention Weeks 4 and 8
  Assessed by self-report ratings of patient-provider connection
Sleep measures | Change from baseline through intervention to 1-week post-intervention and 3-month follow up
  Assessed by self-report ratings of sleep using Pittsburgh Sleep Quality Index
Physiological data (blood pressure, pulse rate) | Change from baseline to 1-week post-intervention and 3-month follow up
  Assessed by blood pressure cuffs in lab
Physiological data (gait) | 1-week post-intervention and 3-month follow up
  Assessed by speed of walking at a normal pace
Perceptual speed and visual attention in daily living | Change from baseline to intervention weeks 4 and 8
  Assessed via a symbol search ambulatory smartphone-based task administered at six timepoints per day, for three days in a row, at baseline and at Intervention weeks 4 and 8
Attentional interference from emotional and social information | 1-week post-intervention
  Emotional Stroop task with negative social, negative non-social, positive social, and positive non-social words
Recall of social and emotional information | 1-week post-intervention
  A social memory task assessing event recall based on event sociality (collective, interpersonal, and individual) and valence (positive and negative)
Selective auditory attention | 1-week post-intervention and 3-month follow-up
  Assessed via a dichotic listening task

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Pawlikowsky, BA, Study Chair — Office of Sponsored Projects, Carnegie Mellon University
Locations (3):
- United States (3):
  - Carnegie Mellon University, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center- Center for Integrative Medicine, Pittsburgh, Pennsylvania
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lindsay EK, Marsland AL, Cole SW, Dutcher JM, Greco CM, Wright AGC, Brown KW, Creswell JD. Mindfulness-Based Stress Reduction Reduces Proinflammatory Gene Regulation But Not Systemic Inflammation Among Older Adults: A Randomized Controlled Trial. Psychosom Med. 2024 Jun 1;86(5):463-472. doi: 10.1097/PSY.0000000000001264. Epub 2023 Nov 17. PMID 37982547
- [Derived] Lindsay EK, Creswell JD, Stern HJ, Greco CM, Dutcher JM, Lipitz S, Walsh CP, Wright AGC, Brown KW, Marsland AL. Mindfulness-Based Stress Reduction Buffers Glucocorticoid Resistance Among Older Adults: A Randomized Controlled Trial. Psychosom Med. 2021 Jul-Aug 01;83(6):641-649. doi: 10.1097/PSY.0000000000000928. PMID 33657083

DOCUMENTS (1):
  • Informed Consent Form (2019-05-31): https://cdn.clinicaltrials.gov/large-docs/00/NCT02888600/ICF_000.pdf